CLINICAL TRIAL: NCT07182474
Title: Turkish Version of the BRIEF-Hammersmith Infant Neurological Examination (HINE) With High-Risk of Infants: A Study of Validity and Reliability
Brief Title: Turkish Version of the BRIEF-Hammersmith Infant Neurological Examination (HINE)
Acronym: BRIEF-HINE
Status: Recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: BRIEF-HINE
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Pediatrics; Neurological Abnormality; Neurodevelopment Outcome
MeSH Terms: conditions — Nervous System Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: High-risk infants referred to the Pediatric Rehabilitation Unit for follow-up will be included. A total of 110±10 high-risk infants will be included in the study, representing 10 times the number of items in the Abstract-HINE version.

SUMMARY:
The American Academy of Pediatrics defines high-risk infants as those with preterm birth, special health care needs, family risk factors, and those at risk of early death. Factors such as premature birth, perinatal asphyxia, hypoxic-ischemic encephalopathy (HIE), periventricular leukomalacia (PVL), intraventricular hemorrhage (IVH), chronic lung disease, seizures, meningitis, hyperbilirubinemia, twin/triplet pregnancy, and intrauterine growth restriction are risk factors that can result in morbidity and mortality in infants. Regular neurological examinations and neuromotor tests are necessary for at-risk infants to identify developmental problems early and to initiate early intervention programs.In developing countries, regular follow-up and early rehabilitation of at-risk infants are not successfully implemented. 5,6 The lengthy test batteries and busy clinics are among the most significant reasons. Therefore, the development and dissemination of shorter, valid, and reliable tests is of great importance. The Hammersmith Neonatal Neurological Examination (HINE), one of the gold standard methods, consists of 26 items and takes 15-20 minutes to administer.Due to the number of items and the duration, it is not frequently used routinely. In response to this clinical need, the HINE short scale was developed in 2024.The aim of the study is to have a Turkish version of the Abstract-HINE test in Turkey and to study its validity and reliability in high-risk infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with high risk of CP: Periventricular hemorrhage, intracranial hemorrhage grade 2, 3, 4, cystic PVL, stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterus), perinatal stroke, perinatal asphyxia, respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD) and infants receiving long-term O₂ support, sepsis due to gram-negative bacteria, necrotizing enterocolitis (NEC), infantile apnea, those with a low 5-minute Apgar score (3 and below), those diagnosed with intrauterine growth retardation, multiple births (twins, triplets), preterm infants with retinopathy of prematurity (ROP), infants with prolonged severe hypoglycemia and hypocalcemia, (small for gestational age (SGA), less than the 3rd percentile) or large for gestational age (large for gestational age (LGA), less than the 97th percentile). (large) babies, babies receiving mechanical ventilation for more than 24 hours, babies born at less than 32 weeks of gestation and weighing less than 1500 grams.

Exclusion Criteria:

* Infants with any known orthopedic, systemic disease or neurological diagnosis other than CP

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with high risk of CP (periventricular hemorrhage, intracranial hemorrhage grade 2, 3, 4, cystic PVL, stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterus), perinatal stroke, perinatal asphyxia, RDS, BPD and infants receiving long-term O₂ support, sepsis due to gram-negative bacteria, NEC, infantile apnea, those with a low 5th minute Apgar score (3 and below), those diagnosed with intrauterine growth retardation, multiple births (twins, triplets), preterm infants with ROP, infants with prolonged severe hypoglycemia and hypocalcemia, infants who are SGA or LGA, infants receiving mechanical ventilation for more than 24 hours, infants born less than 32 weeks of gestation and weighing less than 1500 grams)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The Hammersmith Infant Neurological Examination (HINE) | HINE will be administered to all infants at 3, 6, and 12 months.
  The Hammersmith Infant Neurological Examination (HINE) was developed by Dubowitz and colleagues from a standard neurological examination of newborns. It analyzes the risk of neurological anomalies in preterm and term infants. This test is a prognostic battery for identifying neuromotor disorders in infants between 2 and 24 months postnatally. The HINE scale consists of 37 items divided into three sections: neurological examination, developmental motor milestones, and behavioral status. Administration time is 10-15 minutes. Optimization scores for infants aged 3 to 18 months are based on the frequency distribution of neurological findings in the population in that age group. An item is considered optimal when present in at least 90% of infants. Use of the HINE test's optimality score and cut-off scores for CP at 3, 6, 9, 12, and 24 months provide prognostic information regarding the level of motor development. the HINE will be administered to all infants at 3, 6, and 12 months.
BRIEF-HINE | BRIEF-HINE will be administered to all infants at 3, 6, and 12 months.
  The short form is an 11-item test that takes approximately 5 minutes.This short form includes the 11 subitems of the original HINE, developed by Romeo et al. for use in at-risk infants between 3 and 12 months of age. The item assessment and scoring are the same as the original format, with a 0-3 scale. The total scale score ranges from 0 to 33, with a higher score indicating better neuromotor performance. The test has cut-off values for 3, 6, 9, and 12 months, allowing for categorization of typical/atypical development. The test takes an average of 5 minutes to administer and is well-suited for routine use. The HINE is a valid and reliable test with predictive value, and its Turkish translation has been completed. This study will interpret the cut-off scores for CP.

SECONDARY OUTCOMES:
sosyodemographic form: | Day 1 (at the first time of assessment)
  It will consist of a form that includes prenatal and postnatal risk factors of all infants, demographic information of infants and their parents, and, if available, neurological evaluation, cranial ultrasound (cUS) and Magnetic Resonance Imaging (MRI) results of the infants.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No